CLINICAL TRIAL: NCT05752591
Title: Study of the Hypothalamic-pituitary Dysfuntion in Patients With Diabetes Mellitus
Brief Title: Hypothalamic-pituitary Dysfunction in Diabetes
Acronym: DIAPO
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Marco Bonomi, MD, Professor, Istituto Auxologico Italiano
Other Study IDs: 05C823
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Diabete Mellitus; Hypogonadism; Hypogonadotropic Hypogonadism; Hypergonadotropic Hypogonadism; Central Hypothyroidism
MeSH Terms: conditions — Diabetes Mellitus; Hypogonadism; Hypothyroidism | interventions — Diagnostic Techniques and Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma Whoole Blood DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled patients with DM
  Interventions: Diagnostic Test: Diagnostic testing

INTERVENTIONS:
Diagnostic Test: Diagnostic testing — Blood diagnostic testing for hypothalamic-pituitary-gonadal axis and hypothalamic-pituitary-thyroid axis. In case of gonadal or thyroid dysfunction, genetic testing for known implicated genes

SUMMARY:
Type 2 Diabetes mellitus (T2DM) is a chronic disease with a high prevalence and several comorbidities impacting on public health and society. Among the complications of T2DM it has been showed a high prevalence of hypogonadotropic hypogonadism. Even if hypogonadism is associated to a worse metabolic profile and cardiovascular risk, it is discussed whether and when to treat this potentially reversible form associated to diabetes. In fact, the pathogenic mechanism of this condition in diabetic patients is not fully understood, and its clinical correlates, including the prevalence of other possible associated hypothalamic-pituitary axes dysfunctioning, questioned. The aim of the present study is to assess with an observational, cross sectional study on a large series of type 2 diabetic patients, enrolled consecutively: all the suspected etiologies of this complication in one single evaluation (both acquired and genetic congenital predisposition), its clinical correlates and the real prevalence of the disease using the lastly validated criteria for late onset hypogonadotropic hypogonadism.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years old
* males
* proved diagnosis of T2DM

Exclusion Criteria:

* patients affected with known hypothalamic-pituitary diseases at the enrollment.
* patients affected with severe systemic diseases, fever, chronic inflammatory disorders with PCR > 10 mg/dL
* malnutrition with BMI <17 Kg/m2
* use of glucocorticoids at the enrollment
* poor understanding of spoken and written Italian
* patients affected with known primary diseases of the testes at the enrollment

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Study Population: Cross-sectional, observational study in T2DM patients (minimum 150). The inclusion will be through consecutive enrollment in diabetology clinics.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of Hypogonadism | baseline
  LH, FSH, Testosterone, Estradiol
Genetic predisposition | baseline
  NGS analysis based on the analysis of a customized gene-panel with all known Congenital Hypogonadotropic Hypogonadism genes

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Auxologico Italiano, Milan
  - ASST Fatebenefratelli Sacco, Milan